CLINICAL TRIAL: NCT01676077
Title: International Clinical Outcome Study for Dysferlinopathy
Brief Title: Clinical Outcome Study for Dysferlinopathy
Acronym: Jain COS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Jain Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 85750
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Dysferlinopathy; LGMD2B Now Classified as LGMDR2; Miyoshi Myopathy
Keywords: LGMD2B/ LGMDR9; Miyoshi Myopathy; Dysferlin; Dysferlinopathy; Limb Girdle muscular dystrophy type 2b; Muscular Dystrophy
MeSH Terms: conditions — Dysferlinopathy; Miyoshi myopathy; Limb-girdle muscular dystrophy, type 2B; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA, RNA, Skin fibroblasts, Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with a genetically confirmed dysferlinopathy

SUMMARY:
The "Clinical Outcome Study for Dysferlinopathy" is being performed in centres in Europe (UK- Newcastle; Spain- Barcelona, Sevilla; San Sebastian;Denmark, Copenhagen, Italy- Padova; France- Paris,), USA (Charlotte, NC; Columbus, OH; St.Louis, MO, Stanford CA, Irvine CA and Columbia NY), Chile (Santiago) Japan (Tokyo) and South Korea (Pusan). Oversight is provided by Newcastle upon Tyne Hospitals Trust. Funding for this study is being provided by the Jain Foundation, a non-profit foundation dedicated to finding therapies for dysferlinopathies(LGMD2b/Miyoshi). The aim of this "Clinical Outcome Study" is to determine the clinical outcome measures required for future clinical trials, characterize the disease progression of dysferlinopathy and collect biological samples for the identification of disease markers that are needed to non-invasively monitor the disease during clinical trials. Without this information, effective clinical trials cannot be performed.

This study is recruiting a large number of genetically confirmed dysferlinopathy patients aged 10 years or older, who are ambulant or non-ambulant. The study has reopened for a further two years (COS2). Participants will be assessed at 4 further visits over 2 years via medical, physiotherapy, and MRI/MRS assessments, as well as standard blood tests. Optionally, the participants can donate blood samples and a skin sample for use in the identification of disease markers and other approved research. There is a sub-study running in MRI at selected sites.

DETAILED DESCRIPTION:
Dysferlinopathy represents a rare group of muscular dystrophies, presenting a particular challenge for the definition of natural history and "trial readiness". In the early days after the cloning of the dysferlin gene, several papers described the clinical phenotype over time of collections of patients leading to the recognition of the "core" phenotypes of Miyoshi Myopathy (MM), LGMD2B and the rarer distal myopathy with anterior tibial involvement. Most of these papers dealt with inbred populations with a limited number of mutations represented. Subsequent studies have reported larger numbers of patients with outbred mutations and extended the clinical spectrum to include onset as young as early childhood and as late as old age, with a large group of patients in whom a clear distinction in their pattern of muscle involvement into Miyoshi or LGMD was not possible, with involvement of both the proximal and distal musculature in most patients, especially as the disease progresses. A limitation of all of these studies however is that with few exceptions, again mainly in inbred groups, long-term follow-up data are not presented and data on clinical progression are collected in different ways making precise comparisons between their conclusions difficult. Nonetheless, the studies overall are in agreement that dysferlinopathy is a chronically progressive condition sometimes with periods where there is a plateauing of muscle function, with variable age at wheelchair dependency and probably a low risk of cardiac and respiratory complications compared to other types of muscular dystrophy. Intriguing suggestions from these publications which require more systematic study include the definition of a particularly good level of sporting prowess before the onset of symptoms and the description of a subacute onset with muscle pain and swelling, both features, if better understood, that potentially could help in our understanding of the pathogenesis of the disease.

Recently, two as yet unpublished studies have addressed the topic of charting the natural history of dysferlinopathy more systematically. In a study of 9 genetically confirmed LGMD2B and MM patients studied over 18 months, Isabel Illa and colleagues found a significant decline in muscle strength in a set of muscle groups measured by manual muscle testing, and in knee flexion measured by quantitative muscle testing, accompanied by a detectable deterioration on MRI imaging in biceps femori and tibialis posterior. Maggie Walter and colleagues assessed the natural course of disease and efficacy of deflazacort treatment in 25 patients (between 25 and 63 years of age) with genetically confirmed dysferlinopathy in a double-blind, cross-over trial. During the first year of the study, they assessed the natural course of disease in 6-month intervals, evaluating MRC scores, quantitative strength measurement by hand-held dynamometry (Citec, Groningen, Netherlands), and torque measurement (M3 diagnose system, Fa. Schnell, Germany), Neuromuscular Symptoms Score (NSS), Timed Function Tests (getting up from lying and sitting position, climbing 4 stairs, running 10m), Vignos Scale, Hammersmith Motor Ability Score, and Global Assessment CGI Scale, quality of life SF-36 scale and laboratory parameters (sodium, potassium, creatinine, urea, GOT, GPT, gamma-GT, CK, blood count, ESR, CRP). Medication (placebo or deflazacort in a cross-over design) was only started in the 2nd year of the study. All patients showed a decline in muscle strength over one year, which was reflected in the tests performed.

It is reassuring that from these data we can conclude that it is likely that there will be changes detectable with time in dysferlinopathy that could inform the design of future clinical trials, but the optimal measurements have yet to be defined and mapped in a much larger group of dysferlinopathy patients representing the entire clinical spectrum of this diverse disease group. Extrapolating from the requirements for studies in other types of muscular dystrophies, including the regulatory advice for establishing pivotal trials of therapies in these disorders, these measures would need to include not only measures of muscle strength, but also of function and some degree of patient reported outcomes. The unpublished results of Isabel Illa and colleagues, as well as another small study of MRI in dysferlinopathy, also show some hope for the use of MRI as a measure of change in muscle over time which might be applicable as an outcome measure. Up until now, muscle MRI has been seen more as a tool for delineating the pattern of muscles involved than for monitoring change - the use of MRI for monitoring disease progression in a non-invasive manner is however attracting a lot of current interest, though more study is needed especially in respect of functional correlates and patient relevance.

The frequency of dysferlinopathy provides a further challenge to the collection of natural history data. The relative frequency of different forms of muscular dystrophy depends to a certain extent on the population studied. Dysferlinopathy appears to be a more common cause of LGMD in Southern European populations than in Northern European ones. Founder mutations exist in only a few small communities. There is little doubt that dysferlinopathy is under-diagnosed and, in fact, the clinical diagnostic process by which dysferlinopathy is diagnosed is also variable. Most laboratories still rely on the suggestion of the diagnosis by muscle immunocytochemistry or (more reliably) immunoblotting. Some laboratories carry out protein testing on monocytes as an alternative screening methodology. The gold standard for dysferlinopathy diagnosis has however become DNA testing, with sequencing carried out in a small number of commercial laboratories as well as a series of diagnostic laboratories in Europe and the USA. The Jain Foundation (www.jain-foundation.org) can help guide those who are unsure about their diagnosis through the process of getting a genetic analysis. Please contact Sarah Shira at the Jain Foundation for help with diagnosis at +1 425 882 1492

With the perspective of different approaches to therapy in dysferlinopathy, a clearer definition of the natural history of the disease and the delineation of suitable outcome measures for clinical trials needs to be prioritised. The current protocol builds on existing national and international networks to bring together a critical mass to address the following specific aims:

1. To define the natural history of Dysferlinopathies with respect to age and nature of onset, progression and presence of complications.
2. To determine the most suitable and robust outcomes measures for evaluation of disease progression in patients with Dysferlinopathy at different stages of the disease.
3. To evaluate whether cardiac manifestations are clinically significant in patients with Dysferlinopathy.
4. To explore if sodium MRI could be useful to identify muscle damage on skeletal muscle of patients with Dysferlinopathy

ELIGIBILITY:
Inclusion Criteria:

- Confirmed diagnosis of dysferlinopathy proven by a) two (predicted) pathogenic dysferlin mutations, b) one (predicted) pathogenic dysferlin mutation and absent dysferlin protein on muscle immunoblot, or c) one (predicted) pathogenic dysferlin mutation and dysferlin protein level ≤20% of normal level determined by blood monocyte testing. Mutations will be checked for pathogenicity via the UMD bioinformatics tools and and by checking the literature and mutation /variant databases.

NOTE: Contact Sarah Shira at the Jain Foundation for help with diagnosis at +1 425 882 1492

* Ambulant with or without aids; or full-time wheelchair user, i.e. non-ambulant; with the ratio 2:1 between recruited ambulant and recruited non-ambulant patients.
* All ages ≥ 10 years of age.
* Ability to perform assessments (there will be different assessments for ambulant and non-ambulant patients).
* Ability to attend scheduled investigations.
* Informed consent to participate in the clinical outcome study.

NOTE: Funds are available to cover necessary hotel stays and travel costs to the study centres for the participant and a helper (if needed).

Exclusion Criteria:

* Known current or planned medical or other interventions that might interfere with the possibility to undertake the planned tests.
* Other concomitant pathology that in the view of the investigator would jeopardise the ability to take part in the protocol.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A diagnosis of Limb Girdle Muscular Dystrophy type 2B (LGMD2B/ LGMDR2), Miyoshi myopathy, or any other clinical diagnosis associated with dysferlinopathies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
North Star assessment for limb girdle-type muscular dystrophies (NSAD) | 24 months
  A functional scale that will be used to measure motor performance in individuals with LGMD

CONTACTS AND LOCATIONS:
Overall Officials: Volker Straub, Principal Investigator — Newcastle University; Meredith K James, Principal Investigator — Newcastle University
Locations (16):
- United States (6):
  - UC Irvine, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Neurology & Pathology, Washington University, School of Medicine in St Louis, St Louis, Missouri
  - Columbia University Medical Centre, New York, New York
  - Carolinas Medical Center, Neuroscience & Spine Institute, Dept of Neurology, Charlotte, North Carolina
  - Neuromuscular Center at the Research Institute of Nationwide Children's Hospital, Columbus, Ohio
- Clinica Davila, Santiago, Chile
- Rigshospitalet Neuromusculaer Klinik, Copenhagen, Denmark
- Institut de Myologie, Paris, France
- Department of Neurosciences, University of Padova, Padua, Italy
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan
- Pusan National University Hospital, Busan, South Korea
- Spain (3):
  - Hospital Sant Pau, Neurology Department, Barcelona
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Virgen del Rocio, IBiS, Neurology Department, Seville
- Institute of Translational and Clinical Research, Newcastle University, International Centre for Life, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Moore U, Jacobs M, James MK, Mayhew AG, Fernandez-Torron R, Feng J, Cnaan A, Eagle M, Bettinson K, Rufibach LE, Lofra RM, Blamire AM, Carlier PG, Mittal P, Lowes LP, Alfano L, Rose K, Duong T, Berry KM, Montiel-Morillo E, Pedrosa-Hernandez I, Holsten S, Sanjak M, Ashida A, Sakamoto C, Tateishi T, Yajima H, Canal A, Ollivier G, Decostre V, Mendez JB, Sanchez-Aguilera Praxedes N, Thiele S, Siener C, Shierbecker J, Florence JM, Vandevelde B, DeWolf B, Hutchence M, Gee R, Prugel J, Maron E, Hilsden H, Lochmuller H, Grieben U, Spuler S, Tesi Rocha C, Day JW, Jones KJ, Bharucha-Goebel DX, Salort-Campana E, Harms M, Pestronk A, Krause S, Schreiber-Katz O, Walter MC, Paradas C, Hogrel JY, Stojkovic T, Takeda S, Mori-Yoshimura M, Bravver E, Sparks S, Diaz-Manera J, Bello L, Semplicini C, Pegoraro E, Mendell JR, Bushby K, Straub V; Jain COS Consortium. Assessment of disease progression in dysferlinopathy: A 1-year cohort study. Neurology. 2019 Jan 28;92(5):e461-e474. doi: 10.1212/WNL.0000000000006858. PMID 30626655
- [Derived] Diaz-Manera J, Fernandez-Torron R, LLauger J, James MK, Mayhew A, Smith FE, Moore UR, Blamire AM, Carlier PG, Rufibach L, Mittal P, Eagle M, Jacobs M, Hodgson T, Wallace D, Ward L, Smith M, Stramare R, Rampado A, Sato N, Tamaru T, Harwick B, Rico Gala S, Turk S, Coppenrath EM, Foster G, Bendahan D, Le Fur Y, Fricke ST, Otero H, Foster SL, Peduto A, Sawyer AM, Hilsden H, Lochmuller H, Grieben U, Spuler S, Tesi Rocha C, Day JW, Jones KJ, Bharucha-Goebel DX, Salort-Campana E, Harms M, Pestronk A, Krause S, Schreiber-Katz O, Walter MC, Paradas C, Hogrel JY, Stojkovic T, Takeda S, Mori-Yoshimura M, Bravver E, Sparks S, Bello L, Semplicini C, Pegoraro E, Mendell JR, Bushby K, Straub V; Jain COS Consortium. Muscle MRI in patients with dysferlinopathy: pattern recognition and implications for clinical trials. J Neurol Neurosurg Psychiatry. 2018 Oct;89(10):1071-1081. doi: 10.1136/jnnp-2017-317488. Epub 2018 May 7. PMID 29735511
- [Derived] Moore UR, Jacobs M, Fernandez-Torron R, Jang J, James MK, Mayhew A, Rufibach L, Mittal P, Eagle M, Cnaan A, Carlier PG, Blamire A, Hilsden H, Lochmuller H, Grieben U, Spuler S, Tesi Rocha C, Day JW, Jones KJ, Bharucha-Goebel DX, Salort-Campana E, Harms M, Pestronk A, Krause S, Schreiber-Katz O, Walter MC, Paradas C, Hogrel JY, Stojkovic T, Takeda S, Mori-Yoshimura M, Bravver E, Sparks S, Diaz-Manera J, Bello L, Semplicini C, Pegoraro E, Mendell JR, Bushby K, Straub V. Teenage exercise is associated with earlier symptom onset in dysferlinopathy: a retrospective cohort study. J Neurol Neurosurg Psychiatry. 2018 Nov;89(11):1224-1226. doi: 10.1136/jnnp-2017-317329. Epub 2018 Jan 29. No abstract available. PMID 29378789
- See also: This study is fully funded by the Jain Foundation, a non-profit foundation whose mission is to cure muscular dystrophies caused by dysferlin protein deficiency. — http://www.Jain-foundation.org
- See also: All information for this study can be found on the study website (www.dysferlinoutcomestudy.org), including contact details and participating sites — http://www.dysferlinoutcomestudy.org